CLINICAL TRIAL: NCT04472091
Title: Genicular Artery Embolization for the Treatment of Moderate to Severe Osteoarthritic Knee Pain
Brief Title: Genicular Artery Embolization (GAE) for Osteoarthritic Knee Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Insurance Coverage
Sponsor: Andrew Picel (Other)
Responsible Party: Sponsor-Investigator, Andrew Picel, Assistant Clinical Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 57046; IDE G200111 (Other: FDA)
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Pain Swelling; Knee Arthritis; Arterial Occlusion
Keywords: Knee osteoarthritis; Genicular artery embolization; Geniculate artery embolization
MeSH Terms: conditions — Osteoarthritis, Knee; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Genicular artery embolization (Experimental): Participants will undergo the genicular artery embolization (GAE) procedure for the treatment of moderate to severe knee osteoarthritis. A total of 30 patients will be enrolled in the single treatment arm of the study.
  The study will involve a screening period in which patient eligibility is determined. Once eligibility is confirmed, patients will undergo GAE with HydroPearl® Microspheres (polyethylene glycol microspheres, Terumo Medical, Somerset NJ). Following treatment, patients will undergo follow-up at 1, 6, 12, and 24 months post GAE.
  Interventions: Device: Genicular artery embolization (GAE)

INTERVENTIONS:
Device: Genicular artery embolization (GAE) — Participants will undergo GAE with HydroPearl® Microspheres (polyethylene glycol microspheres, Terumo Medical, Somerset NJ).

SUMMARY:
The objective of this investigation is to evaluate the safety of the geniculate artery embolization (GAE) procedure with HydroPearl® Microspheres in 30 patients with knee pain caused by osteoarthritis with 24 months follow-up. The GAE procedure is an arterial embolization procedure that blocks abnormal blood vessels caused be knee arthritis in order to evaluate the effect on knee pain.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. Age ≥ 40 years
3. Moderate to severe knee pain (VAS >40 mm)
4. Pain refractory to 3 months of conservative treatments, including at least one of the following:

   * a. Anti-inflammatory medications
   * b. Physical therapy
   * c. Intra-articular injections
5. Kellgren-Lawrence radiographic grade 1, 2, or 3 disease
6. MRI features of active synovitis (synovial thickening and/or enhancement on MRI).
7. Ineligibility or refusal of surgical management.
8. Local knee tenderness

Exclusion Criteria:

1. Rheumatoid or infectious arthritis
2. Advanced lower extremity atherosclerosis that would limit selective angiography
3. Local knee infection
4. Prior knee surgery (excluding arthroscopic/meniscal interventions)
5. Uncorrectable coagulopathy (INR>1.8, platelets<50,000/µL)
6. Iodine allergy resulting in anaphylaxis
7. Chronic renal insufficiency (serum creatinine >2 mg/dL)
8. Life expectancy less than 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events | 1 month post GAE
  Adverse events will be evaluated for severity and graded following the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Number of patients with treatment related adverse events | 6 months post GAE
  Adverse events will be evaluated for severity and graded following the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Number of patients with treatment related adverse events | 12 months post GAE
  Adverse events will be evaluated for severity and graded following the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Number of patients with treatment related adverse events | 24 months post GAE
  Adverse events will be evaluated for severity and graded following the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Mean change from baseline pain scores | Baseline to 1 month post GAE
  Pain score measured using visual analogue scale (VAS). The VAS is a numerical scale used to report pain intensity from 0 to 100. Subjects mark the scale with a vertical line to indicate their current pain level. 0 mm represents "no pain" and 100 mm represents "worse possible pain."
Mean change from baseline pain scores | Baseline to 6 months post GAE
  Pain score measured using visual analogue scale (VAS). The VAS is a numerical scale used to report pain intensity from 0 to 100. Subjects mark the scale with a vertical line to indicate their current pain level. 0 mm represents "no pain" and 100 mm represents "worse possible pain."
Mean change from baseline pain scores | Baseline to 12 months post GAE
  Pain score measured using visual analogue scale (VAS). The VAS is a numerical scale used to report pain intensity from 0 to 100. Subjects mark the scale with a vertical line to indicate their current pain level. 0 mm represents "no pain" and 100 mm represents "worse possible pain."
Mean change from baseline pain scores | Baseline 24 months post GAE
  Pain score measured using visual analogue scale (VAS). The VAS is a numerical scale used to report pain intensity from 0 to 100. Subjects mark the scale with a vertical line to indicate their current pain level. 0 mm represents "no pain" and 100 mm represents "worse possible pain."
Mean change from baseline knee function scores | Baseline to 1 month post GAE
  Knee function measured using the Western Ontario and McMaster University Osteoarthritis index (WOMAC) scale. The WOMAC is a 24-question tool that is completed by the patient to evaluate osteoarthritis of the knee, including pain, stiffness, and physical function of the joints. There are 5 items regarding pain, 2 items for stiffness, and 17 items for physical function. Questions are ranked on a 5 point Likert scale. A score of "0" indicates no symptoms and "4" indicates severe symptoms. The individual scores are added and an overall higher score indicates worse symptoms.
Mean change from baseline knee function scores | Baseline to 6 months post GAE
  Knee function measured using the Western Ontario and McMaster University Osteoarthritis index (WOMAC) scale. The WOMAC is a 24-question tool that is completed by the patient to evaluate osteoarthritis of the knee, including pain, stiffness, and physical function of the joints. There are 5 items regarding pain, 2 items for stiffness, and 17 items for physical function. Questions are ranked on a 5 point Likert scale. A score of "0" indicates no symptoms and "4" indicates severe symptoms. The individual scores are added and an overall higher score indicates worse symptoms.
Mean change from baseline knee function scores | Baseline to 12 months post GAE
  Knee function measured using the Western Ontario and McMaster University Osteoarthritis index (WOMAC) scale. The WOMAC is a 24-question tool that is completed by the patient to evaluate osteoarthritis of the knee, including pain, stiffness, and physical function of the joints. There are 5 items regarding pain, 2 items for stiffness, and 17 items for physical function. Questions are ranked on a 5 point Likert scale. A score of "0" indicates no symptoms and "4" indicates severe symptoms. The individual scores are added and an overall higher score indicates worse symptoms.
Mean change from baseline knee function scores | Baseline to 24 months post GAE
  Knee function measured using the Western Ontario and McMaster University Osteoarthritis index (WOMAC) scale. The WOMAC is a 24-question tool that is completed by the patient to evaluate osteoarthritis of the knee, including pain, stiffness, and physical function of the joints. There are 5 items regarding pain, 2 items for stiffness, and 17 items for physical function. Questions are ranked on a 5 point Likert scale. A score of "0" indicates no symptoms and "4" indicates severe symptoms. The individual scores are added and an overall higher score indicates worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Picel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No